CLINICAL TRIAL: NCT03842098
Title: Korean Medicine Patient Registry of Postoperative Therapy for Musculoskeletal Disorders (KPOP-MD): A Study Protocol
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Gachon University Gil Oriental Medical Hospital (Other)
Collaborators: Kyunghee University Medical Center (Other); CHUNG YEON Korean Medicine Hospital (Unknown); Korean medicine hospital of Daejeon University (Unknown); Wonkwang University Iksan Korean Medicine Hospital (Unknown)
Responsible Party: Principal Investigator, Yun-Kyung Song, Principal Investigator, Gachon University Gil Oriental Medical Hospital
Other Study IDs: ISEE_2018_KPOP-MD
Record Dates: First submitted 2019-02-13; First posted 2019-02-15 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: Musculoskeletal Disorders; Korean Medicine Patient Registry; Post-operative Therapy
Keywords: Korean Medicine Patient Registry; Post-operative Therapy; Musculoskeletal Disorders
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Musculoskeletal Disorders patients: Enroll the post operative musculoskeletal disorders patients and follow up their clinic visits and treatment regimen to analyze their utility in healthcare

SUMMARY:
To create an infrastructure that allows for the conduct of prospective, controlled studies comparing the effectiveness of diagnostic and treatment strategies for patients with musculoskeletal disorders after musculoskeletal operations

ELIGIBILITY:
Inclusion Criteria:

* aged 19 and over
* Those who have undergone musculoskeletal related surgery (corresponding to the disease classification code M00-99, S00-99) within 3 years
* voluntary applicant who has no problem with communicate with study associates or a mild cognitive impairment patient who scored higher than 23 points in Korean version of the montreal rating questionnaire with voluntary participation

Exclusion Criteria:

* Participants in other clinical trials
* Those who are unlikely to be adhered to the schedule of clinical studies
* Those who are expected to have difficulty understanding and responding to research questionnaires such as illiteracy, mental and physical weakness

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who suffers from various symptoms after musculoskeletal surgeries
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2022-05-31 (Estimated); Study Completion 2022-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in musculoskeletal pain intensity | At baseline, enrollment after 3/6/9/12 months
  Assessment of musculoskeletal pain intensity by Numeric Rating Scale (NRS)
Change in Disability and estimating quality of life | At baseline, enrollment after 3/6/9/12 months
  Disability and estimating quality of life by Oswestry Disability Index
Change in reduction of pain severity by K-WOMAC | At baseline, enrollment after 3/6/9/12 months
  Assessment of pain severity by K-WOMAC
Change in Pain and disability of the shoulder by SPADI questionnaire | At baseline, enrollment after 3/6/9/12 months
  Assessment of Pain and disability of the shoulder by SPADI questionnaire
Change in current health status | At baseline, enrollment after 3/6/9/12 months
  The health status will be observed with the Euroqol (EQ-5D-5L) questionnaire.
Change in Severity assessment of any symptoms other than pain | At baseline, enrollment after 3/6/9/12 months
  Severity assessment of any symptoms other than pain by Numeric Rating Scale (NRS)

CONTACTS AND LOCATIONS:
Overall Officials: Yun-Kyung Song, PhD, Principal Investigator — Gachon University Gil Oriental Medical Hospital
Locations (1):
- Gachon universiry affiliated Gil oriental medicine hospital, Incheon, South Korea

IPD SHARING:
Plan to Share IPD: No
denial from study associates